CLINICAL TRIAL: NCT04277299
Title: Intelligent Customer-driven Solution for Children and Their Parents Undergoing Children´s Day Surgery
Brief Title: Intelligent Customer-driven Solution for Children and Their Parents Undergoing Day Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: VTT Technical Research Centre of Finland (Other); Hospital District of Helsinki and Uusimaa (Other); Tampere University (Other); Buddy Healthcare Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HUS180/2020
Record Dates: First submitted 2020-02-10; First posted 2020-02-20 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Tonsillitis; Herniorrhaphies; Surgery; Children; Parents
MeSH Terms: conditions — Tonsillitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The participants in the intervention group will receive the routine care plus the ICory-Solution which is the surgical pathway currently practiced in the study hospital. The ICory-Solution has two components: (1) the Buddy Healthcare mobile app (BuddyCare) that provides a comprehensive day-by-day perioperative guide for parents regarding their child's surgery with an interface for health care professionals to monitor parents' and their children's needs as well as communicate with them. (2) The Triumf Health mobile game app that provides emotional support and distraction to children.
  Interventions: Device: IcorySolution
- Control group (No Intervention): Children in the control group will receive routine care provided by the hospital which consists of normal doctor consultant, preoperative preparation, and postoperative care. Parents in this group will receive BuddyCare mobile app which is supposed to be as a normal routine in this hospital.

INTERVENTIONS:
Device: IcorySolution — The ICory-solution programme is designed to be a self-guided and healthcare professional-led. Participants will have access to BuddyCare for parents and Triumf Health from time of recruitment till 2 weeks after surgery. The healthcare professional have received face-to-face training on how to use the BuddyCare dashboard and BuddyCare has been in the hospital in earlier studies.The Buddy Healthcare mobile app (BuddyCare) that provides a comprehensive day-by-day perioperative guide for parents regarding their child's surgery with an interface for health care professionals to monitor parents' and their children's needs as well as communicate with them. (2) The Triumf Health mobile game app that provides emotional support, games and distraction to children and a virtual tour to the hospital before children´s operation.
  Arms: Intervention group

SUMMARY:
This research aims to evaluate the effectiveness of web-based mobile intervention (Icory -Solution) developed to pediatric patients and their parents in the pathway of outpatient surgery treatment in pre-intra- and postoperative setting: (1) Examine the effectiveness of the intervention on children's preoperative anxiety and fear, and postoperative pain (2) examine the effectiveness of the intervention on parental anxiety and satisfaction in children´s care path and (3) examine the experiences of the gamification in children in the intervention group.

DETAILED DESCRIPTION:
Children and their families are entitled to know what is going to happen to them before undergoing day surgery and information must be based on the child's age and understanding. It is important to help children to cope with any upcoming surgery because the more anxious and fear they are, the more pain they experience after the day surgery. Digital gaming solutions could help families and children to be better oriented to the coming treatment. Icory -solution is a digital pathway for children and family and it contains a virtual tour to hospital and distraction games for children. The information on the application is aligned with the patient's individual needs based on the type of surgery and requirements.

ELIGIBILITY:
Inclusion Criteria:

* Age between 7-12 years old
* Is scheduled for an elective day surgery
* Is able to speak, and read in Finnish
* Is accompanied by their parents (either mother or father or both) during the perioperative period
* Has access to smart phone/tablet (own or rent from the project)

Exclusion Criteria:

* Cognitive and learning disabilities identified from the medical record
* A chronic illness and/or pain that required special medical care

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
mYPAS | mYPAS will be assessed at the baseline:(1)at the hospital on the day before the operation when nurse meets the child, and will assess changes between baseline and (2) before the induction and (3) one hour after operation when the child is awakening
  Children's preoperative anxiety: Modified Yale Preoperative Anxiety Scale - (mYPAS-) Modified Yale Preoperative Anxiety Scale ( Kain et al 1997) will be used to measure the preoperative anxiety levels of the children right before the operation. It is a 4-item scale (activity, vocalization, emotional expressivity, state of apparent arousal) and it is filled in via observation. The total score ranges from 23 to 100. Higher scores mean higher levels of anxiety. A score of 31 and above would indicate high-anxiety.

SECONDARY OUTCOMES:
CPMAS | CPMAS will be assessed (1) one day before the operation at home, and will be assessed changes between baseline and (2) at the hospital before the operation and (3) before the induction and (4) days 1 and (5) 7 after the operation
  Children's Perioperative Multidimensional Anxiety Scale (CPMAS) developed by Chow et al. (2015) is a simple, age-appropriate self-report measure of pediatric perioperative anxiety and fear in busy hospital settings. The CPMAS is a visual analog scale composed of 5 items, each of which is scored from 0-100.
Children´s postoperative pain | Children's postoperative pain will be measured at baseline (1) right after the operation and will be assessed changes between baseline (2) 24 hours,(3) days 3 and (4) 7 post-surgery
  VAS - The visual analogue scale (VAS) is a psychometric response scale to measure children´s postoperative pain. The scores range from 0-100 (Abu-Saad 1984) with a higher score means greater pain.
STAI- Y | Parents' preoperative anxiety will be assessed at baseline (1) at home on the day before the operation and will assess changes between baseline on the surgery day and (2) after the operation and (3) 24 hours after children´s day surgery
  Parental anxiety Parental anxiety STAI- Y form will be used to measure parental anxiety using the State-Trait Anxiety Inventory (STAI-Y) which is a psychological inventory based on a 4-point Likert scale and consists of 20 questions on a self-report basis (Copyright © 1983 by Charles D. Spielberger)
Parental satisfaction: VAS | Parents' satisfaction on children´s day care path will be assessed at baseline (1) at home on the day and (2) on the surgery day after the operation and (3) 24 hours after children´s day surgery
  Parental satisfaction Satisfaction VAS (Reported satisfaction level by visual analog scales 1-10) 0 not at all satisfied 10 very satisfied
GAMEFULQUEST | Gamefulquest will be assessed 1 week after the operation
  Gamefulquest -instrument (Högberg et al. 2019) is a questionnaire for children in the intervention group to measure children´s experience playing the Triumf game. Gamefulquest is a 7-point Likert scale (1 totally disagree - 7 totally agree) concerning children's experience of playing the game in track record, immersion, challenge, playfulness and communal experience

CONTACTS AND LOCATIONS:
Overall Officials: Pekka Lahdenne, Principal Investigator — New Children´s Hospital
Locations (1):
- New Children´s Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
Due to GDPR in Finland, we doesn't plan to share data to public

REFERENCES:
- [Background] Chow CHT, Van Lieshout RJ, Schmidt LA, Buckley N. Tablet-Based Intervention for Reducing Children's Preoperative Anxiety: A Pilot Study. J Dev Behav Pediatr. 2017 Jul/Aug;38(6):409-416. doi: 10.1097/DBP.0000000000000454. PMID 28661955
- [Background] Abu-Saad H. Assessing children's responses to pain. Pain. 1984 Jun;19(2):163-71. doi: 10.1016/0304-3959(84)90836-4. PMID 6462728
- [Background] Högberg, J., Hamari, J., & Wästlund, E. (2019). Gameful Experience Questionnaire (GAMEFULQUEST): an instrument for measuring the perceived gamefulness of system use. User Modeling and User-Adapted Interaction, 1-42.
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Spielberger CD (1983) Manual for the State-Trait Anxiety Inventory (STAI: Form Y). Palo Alto, CA: Consulting Psychologists Press, 1983:4-26
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820
- [Background] Kerimoglu B, Neuman A, Paul J, Stefanov DG, Twersky R. Anesthesia induction using video glasses as a distraction tool for the management of preoperative anxiety in children. Anesth Analg. 2013 Dec;117(6):1373-9. doi: 10.1213/ANE.0b013e3182a8c18f. PMID 24257388
- [Background] Kim H, Jung SM, Yu H, Park SJ. Video Distraction and Parental Presence for the Management of Preoperative Anxiety and Postoperative Behavioral Disturbance in Children: A Randomized Controlled Trial. Anesth Analg. 2015 Sep;121(3):778-784. doi: 10.1213/ANE.0000000000000839. PMID 26176357
- [Background] Lee JH, Jung HK, Lee GG, Kim HY, Park SG, Woo SC. Effect of behavioral intervention using smartphone application for preoperative anxiety in pediatric patients. Korean J Anesthesiol. 2013 Dec;65(6):508-18. doi: 10.4097/kjae.2013.65.6.508. Epub 2013 Dec 26. PMID 24427456
- [Background] Liguori S, Stacchini M, Ciofi D, Olivini N, Bisogni S, Festini F. Effectiveness of an App for Reducing Preoperative Anxiety in Children: A Randomized Clinical Trial. JAMA Pediatr. 2016 Aug 1;170(8):e160533. doi: 10.1001/jamapediatrics.2016.0533. Epub 2016 Aug 1. PMID 27294708
- [Background] Marechal C, Berthiller J, Tosetti S, Cogniat B, Desombres H, Bouvet L, Kassai B, Chassard D, de Queiroz Siqueira M. Children and parental anxiolysis in paediatric ambulatory surgery: a randomized controlled study comparing 0.3 mg kg-1 midazolam to tablet computer based interactive distraction. Br J Anaesth. 2017 Feb;118(2):247-253. doi: 10.1093/bja/aew436. PMID 28100529
- [Background] Messeri A, Caprilli S, Busoni P. Anaesthesia induction in children: a psychological evaluation of the efficiency of parents' presence. Paediatr Anaesth. 2004 Jul;14(7):551-6. doi: 10.1111/j.1460-9592.2004.01258.x. PMID 15200651
- [Background] Moher D, Schulz KF, Altman DG. The CONSORT statement: revised recommendations for improving the quality of reports of parallel-group randomised trials. Lancet. 2001 Apr 14;357(9263):1191-4. PMID 11323066
- [Background] Pope N, Tallon M, McConigley R, Leslie G, Wilson S. Experiences of acute pain in children who present to a healthcare facility for treatment: a systematic review of qualitative evidence. JBI Database System Rev Implement Rep. 2017 Jun;15(6):1612-1644. doi: 10.11124/JBISRIR-2016-003029. PMID 28628521
- [Background] Niemelä, R., Pikkarainen, M., Ervasti, M., & Reponen, J. (2019). The change of pediatric surgery practice due to the emergence of connected health technologies. Technological Forecasting and Social Change, 146, 352-365. https://doi.org/10.1016/j.techfore.2019.06.001
- [Background] Seiden SC, McMullan S, Sequera-Ramos L, De Oliveira GS Jr, Roth A, Rosenblatt A, Jesdale BM, Suresh S. Tablet-based Interactive Distraction (TBID) vs oral midazolam to minimize perioperative anxiety in pediatric patients: a noninferiority randomized trial. Paediatr Anaesth. 2014 Dec;24(12):1217-23. doi: 10.1111/pan.12475. Epub 2014 Jul 17. PMID 25040433
- [Background] Stewart B, Cazzell MA, Pearcy T. Single-Blinded Randomized Controlled Study on Use of Interactive Distraction Versus Oral Midazolam to Reduce Pediatric Preoperative Anxiety, Emergence Delirium, and Postanesthesia Length of Stay. J Perianesth Nurs. 2019 Jun;34(3):567-575. doi: 10.1016/j.jopan.2018.08.004. Epub 2018 Nov 7. PMID 30413359
- [Derived] Rantala A, Vuorinen AL, Koivisto J, Simila H, Helve O, Lahdenne P, Pikkarainen M, Haljas K, Polkki T. A gamified mobile health intervention for children in day surgery care: Protocol for a randomized controlled trial. Nurs Open. 2022 Mar;9(2):1465-1476. doi: 10.1002/nop2.1143. Epub 2021 Dec 2. PMID 34859602